CLINICAL TRIAL: NCT06356428
Title: Psychometric Properties and Cross-cultural Adaptation of the Turkish Version of Physcian Attitudes Toward Cardiac Rehabilitation and Referral Scale-Revised (PACRR-R)
Status: Recruiting | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Haluk Tekerlek, Research assistant, PhD, Karamanoğlu Mehmetbey University
Other Study IDs: KARYÖN-DR
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Physician's Role

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physcian Attitudes toward Cardiac Rehabilitation and Referral Scale-Revised (PACRR-R) — The PACRR comprises 20 items and 1 open ended item to assess physicians' attitudes and beliefs about CR and referral (includes instructions for scale completion to respondents). Response options were 1 = strongly disagree, 2 = agree, 3 = neutral, 4 = agree, and 5 = strongly agree. Five (5) items are reverse-scored to mitigate acquiescence bias (denoted with *), such that higher scores reflect more positive atti- tudes toward CR and referral. A mean score is computed for the total (where at least 80% of items were completed; i.e., 15/19) scale and subscales.

SUMMARY:
Research has reported that the reasons for low implementation of CR are multifactorial at the health system, physician and patient levels. It has also been found that patients are more likely to initiate CR if physicians strongly and positively promote the importance of CR participation. Unfortunately, there are insufficient and ineffective data on CR, referral to CR and both clinical and cost-effectiveness outcomes of CR in Turkey. In this context, it is important to examine more objectively from the perspective of physicians who play a key role in referring patients to CR. However, in our country, there is no relatively objective measurement tool to evaluate physicians' attitudes towards CR. Therefore, this study aims to adapt the original "Physician Attitudes towards Cardiac Rehabilitation and Referral Scale-Revised (PACRR-R)" into Turkish and to examine its psychometric properties.

ELIGIBILITY:
Inclusion Criteria:

* To be a physician,
* Providing active service in patient diagnosis and treatment

Exclusion Criteria:

* Not providing active service in patient diagnosis and treatment despite being a physician (administrative position, etc.).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of the study is physicians. The sample was physicians who volunteered to participate in the study, to whom the study could be announced/notified, and who provided active service in patient diagnosis and treatment. In the literature, it is stated that the number of individuals to be included in the study in order to achieve meaningful and valid results in the scale development process is at least 5 times the number of items in the scale and ideally 10 times. In our study, the number of individuals to be included in the study to test the validity of the scale was planned to be at least 100 individuals (PACRR-R consists of 20 items). In order to examine the test-retest reliability of the scale, it was planned to reapply the scale to at least 25% of the individuals in the sample.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-13 (Estimated); Primary Completion 2025-05-13 (Estimated); Study Completion 2025-08-13 (Estimated)

PRIMARY OUTCOMES:
Physician Attitudes toward Cardiac Rehabilitation and Referral (PACRR)-Revised Scale Score | 10-15 minutes
  The Physician Attitudes toward Cardiac Rehabilitation and Referral (PACRR)-Revised Scale comprises 20 items to assess physicians' attitudes and beliefs about CR and referral. Response options were 1 = strongly disagree, 2 = agree, 3 = neutral, 4 = agree, and 5 = strongly agree. Five (5) items are reverse-scored to mitigate acquiescence bias (denoted with *), such that higher scores reflect more positive attitudes toward CR and referral. A mean score is computed for the total (where at least 80% of items were completed; i.e., 15/19) scale and subscales. A final open-ended item asks physicians to list the most important factors that influence their decision to refer a patient to CR.

CONTACTS AND LOCATIONS:
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided